CLINICAL TRIAL: NCT07390526
Title: The Effect of Perceived Social Support Levels on Life Satisfaction and Social Participation in Adult Stroke Patients
Brief Title: Perceived Social Support in Adult Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Seda Nur Kemer, Principal investigator, PT, PhD, Ondokuz Mayıs University
Other Study IDs: 2025/104
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Healthy Control
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke Patients
- Healthy control

SUMMARY:
Given the limited evidence in the literature regarding the effect of perceived social support on life satisfaction and social participation in adults with stroke, this study aimed to investigate the effect of perceived social support on these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Score ≥24 on the Standardized Mini-Mental Test (SMMT) or Mini-Mental State Examination-Education (MMSE-E)
* Proficiency in Turkish
* Voluntary participation
* For the stroke group: clinical diagnosis of stroke at least 3 months prior to enrollment
* For the stroke group: certified disability rate of at least 20%

Exclusion Criteria:

* Unwillingness to participate
* Presence of major neurological disorders other than stroke
* Orthopedic disorders affecting the musculoskeletal system
* Rheumatic disorders affecting the musculoskeletal system
* For the stroke group: history of multiple strokes
* For the stroke group: presence of bilateral hemiplegia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients and age-matched healthy controls
Sampling Method: Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-02-21 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Mini Mental State Examination | Baseline
  Cognitive function was assessed using the Mini-Mental State Examination (MMSE), a 30-point scale ranging from 0 to 30, where higher scores indicate better cognitive function.
Brunnstrom Stages of Hemiplegic Recovery | Baseline
  Motor recovery was assessed using the Brunnstrom Stages of Hemiplegic Recovery for the upper extremity, hand, and lower extremity, which classify motor function into six sequential stages (Stage I-VI), with higher stages indicating better motor recovery.
The Satisfaction with Life Scale | Baseline
  Life satisfaction was assessed using the Satisfaction with Life Scale (SWLS), a five-item scale with total scores ranging from 5 to 35, where higher scores indicate greater life satisfaction.
Short Form-36 Health Survey (SF-36) | Baseline
  Health-related quality of life was assessed using the Short Form Health Survey (SF-36), which yields scores ranging from 0 to 100 for each domain, with higher scores indicating better health-related quality of life.
Multidimensional Scale of Perceived Social Support | Baseline
  Perceived social support was assessed using the Multidimensional Scale of Perceived Social Support (MSPSS), a 12-item scale with total scores ranging from 12 to 84, where higher scores indicate greater perceived social support.
Modified Mini-Mental State Examination for Illiterate Individuals | Baseline
  Cognitive function was assessed using the Modified Mini-Mental State Examination (3MS), which yields scores ranging from 0 to 100, with higher scores indicating better cognitive function.

IPD SHARING:
Plan to Share IPD: No